CLINICAL TRIAL: NCT01538732
Title: Single-Center, Prospective, Open Label, Single-arm Pilot Study Investigating the Efficacy and Safety of Alitretinoin in Patients Suffering From Severe Mucosal Lichen Planus.
Brief Title: Lichen Planus Mucosae at USZ, Efficacy of Oral Alitretinoin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LISZT-2012
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Lichen Planus (LP)
MeSH Terms: conditions — Lichen Planus | interventions — Alitretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: alitretinoin — 30mg capsules (Alitretinoin)will be taken peroral once daily with a meal. Study treatment will be given for a total duration of up to 24 weeks

SUMMARY:
This is a single center, prospective, open label, single arm, investigator initiated pilot study investigating the effect of alitretinoin on severe lichen planus with mucosal manifestations. The target population comprises patients with MLP for at least 3 months, with or without LP lesions on other areas of the skin, who are refractory to topical therapy and standard skin care, and who are otherwise in good health. Patients will be recruited at the outpatient clinic of the dermatology department, University hospital Zurich.The planned duration of the study is 2 years. A total of 20 patients will be included. Patients who meet enrolment criteria will receive 30mg alitretinoin, given orally as gelatin capsules, once daily for 24 weeks. Dose interruptions are permitted in response to adverse effects, consistent with use of retinoids and the product label.

Most clinical evaluations will be performed every 4 weeks. A safety follow-up visit is planned 4 weeks after the end of treatment. Further follow-up visits will be conducted 16 and 24 weeks after end of treatment in those patients meeting the primary endpoint

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria

* Aged 18 to 75 years
* MLP for at least 3 months
* Disease activity according to Escudier score of 10 points or greater or erosive lesion of any score
* Refractory to standard topical therapy
* Consensus to a 2 weeks wash-out period of topical steroids before starting study treatment

Exclusion criteria

* Unable to comply with the requirements of the study
* Pregnant or lactating women
* Female patients of childbearing potential who cannot use or will not commit to using two effective forms of contraception simultaneously under supervision of the investigator or a gynecologist
* Active hepatitis and/or vaccination against hepatitis A/B during the last 4 weeks
* Adequate control of the disease by standard topical therapy and standard topical corticosteroid therapy
* Known hypersensitivity to other retinoids or vitamin A derivatives, or to any study medication component
* Patients treated with any of the following treatments 4 weeks before the start of study treatment:

  1. systemic drugs: corticosteroids, immunosuppressants, methotrexate
  2. phototherapy
* Treatment with any systemic or topical retinoids within 1 year or 1 month, respectively, before start of study treatment or treatment with systemic retinoids for treatment for MLP at any time
* coexistence of any serious medical condition which, in the opinion of the investigator, may interfere with the safety of the patient, including

  1. hepatic insufficiency (alanine aminotransferase and /or aspartate aminotransferase values > 2.5 x ULN)
  2. severe renal failure
  3. uncontrolled hypertriglyceridemia (triglycerides >150 % of the upper limit of normal),
  4. uncontrolled hypercholesterolemia (cholesterol or low density lipoprotein (LDL) cholesterol values > 1.5 x ULN
  5. Patients with cardiovascular risk factors that would exclude a starting dose of 30 mg of alitretinoin
  6. Uncontrolled hypothyroidism
  7. Hypervitaminosis A
  8. Active major psychiatric disorder including depression and suicidal ideation
* Concomitant medications such as systemic tetracyclines, CYP3A4 inhibitors such as ketoconazole, Vitamin A or St. John's Wort within 1 week, or receiving systemic itraconazole within 2 weeks, before start of study treatment
* Trial participation within 2 months before start of study treatment (3 months for biologics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of alitretinoin (Toctino®) based on the Escudier score of oral lesions at baseline and after 24 weeks of treatment. | 6 months
  The primary objective is to determine the efficacy of alitretinoin (Toctino®) in reducing signs and symptoms of severe mucosal lichen planus with respect to the proportion of responders based on the, Escudier score of oral lesions at baseline and after 24 weeks of treatment or at the latest assessment for patients who withdrew prematurely (Last Observation Carried Forward, LOCF). Response is defined as a 50 % reduction in the total Escudier score compared to the baseline values.

SECONDARY OUTCOMES:
Assess the efficacy of alitretinoin over time in reduction of signs (e.g. ulcerations) or symptoms (e.g. pruritus), using VAS for pruritus and pain and OHIP | 6 months
Assess the time to response (time to 50 % reduction in the total Escudier score) | 6 months
Assess oral mucosal changes regarding inflammation and erosions, at treatment end compared to baseline using Escudier | 6 months
Assess the number/distribution of extramucosal skin lesions (papules) of LP at treatment end compared to baseline | 6 months
Assess, if applicable, the inflammatory infiltrate in mucosa and skin before and during alitretinoin therapy determined by histopathology taken before and 4 weeks after initiation of study treatment. | 4 weeks
Determine the relapse rate (relapse is defined as Escudier score or number of extramucosal papules increasing back to > 75% of baseline) within 24 week follow-up | 6 months
Assess safety of alitretinoin in mucosal lichen planus for the body as a whole | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, Prof. MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Division of Dermatology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Kunz M, Urosevic-Maiwald M, Goldinger SM, Frauchiger AL, Dreier J, Belloni B, Mangana J, Jenni D, Dippel M, Cozzio A, Guenova E, Kamarachev J, French LE, Dummer R. Efficacy and safety of oral alitretinoin in severe oral lichen planus--results of a prospective pilot study. J Eur Acad Dermatol Venereol. 2016 Feb;30(2):293-8. doi: 10.1111/jdv.13444. Epub 2015 Oct 27. PMID 26507685